CLINICAL TRIAL: NCT07147439
Title: Turkish Validity and Reliability of the Appetite Loss in Older Adults With and Without Cognitive Impairment (ALOC) Screening Scale
Brief Title: Turkish Validation of the ALOC Screening Scale in Older Adults
Acronym: ALOC
Status: Not yet recruiting | Type: Observational
Sponsor: Toros University (Other)
Responsible Party: Principal Investigator, Betül Gülşen, Assoc. Prof., Toros University
Other Study IDs: 21.04.2025-04-73
Record Dates: First submitted 2025-08-21; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Elderly (People Aged 65 or More); With or Without Cognitive Impairment
Keywords: Elderly; ALOC; SNAQ; TURKISH VALIDITY AND RELIABILITY

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elderly with or without cognitive impairment: The data collection process of the research will be carried out in four different nursing homes in Mersin province. For this study, a total of 300 older adults will be reached. Within the scope of the research, one-on-one interviews will be conducted with elderly individuals staying in these nursing homes and "scale questions planned to be adapted into Turkish" and "descriptive information forms" will be used.
- The data collection process of the research will be carried out in four different nursing homes.: Within the scope of the research, one-on-one interviews will be conducted with elderly individuals staying in these nursing homes and "scale questions planned to be adapted into Turkish" and "descriptive information forms" will be used.

SUMMARY:
As the elderly population increases, health problems related to aging are also increasing. Loss of appetite negatively affects public health by causing malnutrition and related health problems in elderly individuals. Loss of appetite is a common problem in older adults, both in individuals with and without cognitive impairment. This can lead to serious health problems such as malnutrition, weight loss, muscle loss, weakening of the immune system and decreased quality of life. Cognitive disorders such as Alzheimer's and dementia can trigger loss of appetite, or loss of appetite can be a symptom of these disorders. Factors such as metabolic changes during the aging process, decreased sense of taste and smell, loneliness and depression contribute to loss of appetite. However, there is no valid and reliable scale in Turkey for the early diagnosis and assessment of loss of appetite. A scale being valid and reliable means that it can measure the concept it is intended to measure accurately and consistently. The aim of this study was to determine the validity and reliability of the Turkish version of the Loss of Appetite Scale in older adults with and without cognitive impairment .

DETAILED DESCRIPTION:
Appetite plays an important role in food intake, and anorexia is recognized as an important factor in the development of malnutrition. Anorexia is reported by up to 27% of community-dwelling older adults and is associated with adverse health outcomes such as disability and death. The relationship between appetite and malnutrition is primarily influenced by diet, and it can be assumed that people with anorexia consume less food and make less positive food choices. Age-related changes in gut hormones may play a role in anorexia of aging. Anorexia of aging describes the age-related decline in appetite and food intake experienced later in life. Loss of appetite affects more than 30% of community-dwelling older adults and up to 60% of hospitalized older adults . Anorexia of age has been suggested to be strongly associated with undernutrition, which is associated with sarcopenia, frailty and mortality. This results in a significant increase in healthcare utilization. Annual health and social care costs are estimated to be 3 times higher for undernourished older adults compared to those who are adequately nourished. With an ageing world population, undernutrition in old age poses a challenging problem for current and future healthcare services.

Although anorexia of old age is a common clinical dilemma in hospitals, it is often not routinely assessed and diagnosed. There are several reasons for this, firstly, the lack of consensus on its assessment using different scales or proxy measures such as food intake or weight, which blurs the line between anorexia and malnutrition. However, the Council on Nutritional Appetite Questionnaire (CNAQ) and particularly its shortened version, the 4-question Simplified Nutritional Appetite Questionnaire (SNAQ), which gives a score out of 20 (<14 suggests anorexia), are increasingly used in clinical research settings and may therefore be a suitable tool for use in hospital settings. In addition, the lack of knowledge about the effects of anorexia of old age on health outcomes and the lack of evidence on management strategies to address when the problem is identified also hinder progress in routine clinical practice.

In the hospital setting, the factors most associated with appetite are physical factors, usually related to eating. In this context, the impact of oral health is quite striking. In a study conducted on rehabilitation patients in Japan, anorexia (defined as a SNAQ score ≤14) was found to be 2.7 times more associated with poor oral health using the Oral Health Assessment Tool (OHAT). The OHAT assesses the condition of teeth, mucous membranes and saliva with different subcategories. In this study, subcategories such as poor oral hygiene and the use of dentures were associated with anorexia. These findings are consistent with the results of Donini et al., who observed that older adults with anorexia in hospitals and rehabilitation centers in Italy had fewer natural teeth (5±7 vs. 10±11). Anorexia was defined as the inability to consume at least 50% of a standard meal, without physical factors limiting eating, and lasting for more than three days. In the same study, problems such as chewing difficulty and dysphagia (difficulty swallowing) were also reported to be associated with anorexia. Similarly, this association was observed in older adults presenting to the emergency department in Denmark using a SNAQ score <14. In addition, another study conducted in Japan revealed that the use of texture-modified diets (defined as International Dysphagia Diet Standardization Initiative (IDDSI) levels 3-5) increased the risk of anorexia (odds ratio 3.443).

Other physical factors that affect appetite in the hospital setting include pain, constipation, low cognitive function, and polypharmacy (use of ≥5 different medications). Inflammation and inflammatory cytokines also play an important role in anorexia. Observational studies have shown an association between high C-reactive protein (CRP) levels and reduced food intake in elderly patients In a study conducted in Germany on elderly patients, the relationship between appetite (measured using the SNAQ questionnaire and the Edmonton Symptom Assessment System (ESAS)) and inflammatory markers was investigated. A significant association was found between CRP levels and appetite, independent of the presence of infection or chronic inflammatory disease, age and gender. Focusing on inflammatory cytokines, changes in IL-6 and IL-18 were associated with ESAS-appetite, while IL-10 and IL-33 were associated with SNAQ-appetite. In particular, changes in IL-18 levels were identified as the main predictors of changes in ESAS-appetite.

Mood is closely related to appetite levels in both men and women. In hospitalized elderly individuals, low mood assessed using the Geriatric Depression Scale Short Form (GDS-15) is associated with poor appetite measured with the SNAQ. However, these low mood states do not reach the threshold required to diagnose depression (median score is 4 out of 15, depression threshold is ≥5), increasing the risk of being missed in the clinic. Low mood is linked to hedonic appetite, which includes the reward and pleasure dimension of eating, and affects the desire to eat. However, the lack of research examining the effects of acute illness and inflammation on mood and appetite requires further work in this area.

Physical activity is also an important factor associated with appetite. A study of elderly patients in the United Kingdom showed that higher levels of physical activity prior to hospital admission were associated with better appetite (measured with the SNAQ 13), using the Physical Activity Scale for the Elderly (PASE).

Physical activity is thought to help a person consume the amount of food they need by regulating appetite signals. However, changes in appetite signals during aging may make this relationship more complex. Physical activity levels decrease significantly during hospitalization, which can have an impact on appetite. More research is needed in this area.

The co-creation of food and dietary recommendations has been well received across a range of nutrients including fibre and protein. However, it must be acknowledged that there are marked individual differences in social gradients and health across older adult groups and this is not always represented in current literature. Raising awareness of dietary and nutritional requirements in this population group is still needed and much can be gained by consulting older adults when exploring solutions.

Age-related changes in the complex appetite regulation system, referred to as anorexia of aging, predispose older adults to reduced food intake and may lead to malnutrition if additional risk factors such as health or social problems occur. Consequently, malnutrition is common in the elderly population, especially in those living in institutions. Despite the availability of effective interventions, malnutrition prevention and treatment still do not receive the attention they deserve. As an important first step towards better awareness, malnutrition screening should become a mandatory part of comprehensive geriatric assessment. Furthermore, practical local guidelines should be implemented in all geriatric hospital wards and nursing homes to improve nutritional care in daily routine.

Cognitive disorders can affect the areas of the brain that regulate appetite, causing loss of appetite. The hypothalamus, in particular, is an important center that controls appetite and hunger signals. In neurodegenerative disorders such as Alzheimer's disease, damage to neurons in the hypothalamus can lead to loss of appetite. In addition, reduced senses of taste and smell in individuals with cognitive impairment can also negatively affect the desire to eat.

Appetite loss can cause serious health problems in elderly individuals with cognitive diseases. In addition to physical problems such as malnutrition, muscle loss, weakened immune system, and susceptibility to infections, psychological effects such as depression and social isolation can also be observed. Therefore, early detection and management of appetite loss is of great importance. Management of appetite loss in elderly individuals with cognitive diseases requires a multidisciplinary approach. Nutritional support, behavioral interventions, and pharmacological treatments are important components of this process. For example, consumption of high-calorie and nutrient-rich foods can help meet the energy needs of individuals. In addition, improving the eating environment and increasing social interactions can also positively affect appetite. Appetite loss in elderly individuals with cognitive diseases is an important problem that negatively affects both physical and psychological health. Early detection and effective management of this condition are critical to improving the quality of life of individuals. In future studies, it is recommended to develop innovative strategies to prevent appetite loss.

The aim of this study was to determine the validity and reliability of the Turkish version of the Loss of Appetite Scale in older adults with and without cognitive impairment.

H1: Loss of appetite scale in older adults with and without cognitive impairment, which will be adapted into Turkish, is a valid measurement tool.

H2: Loss of appetite scale in older adults with and without cognitive impairment, which will be adapted into Turkish, is a reliable measurement tool.

ELIGIBILITY:
Inclusion Criteria:

* Elderly over 65 years, with or without cognitive impairment

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The data collection process of the research will be carried out in four different nursing homes in Mersin province, namely Mersin Aid and Kindness Foundation Retirement Home, Mersin Sevgi Bağı Retirement Home, Private Mersin Bahar Retirement Home and Private Alya Elderly Care Center and Retirement Home. The interviews will be conducted in an atmosphere suitable for the participants to express themselves in a comfortable and safe environment. In addition, within the framework of ethical rules, the participants will be included in the research on a voluntary basis and the confidentiality of their information will be protected. The collected data will be analyzed in line with the purpose of the research and the results will be evaluated.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Validity and Reliability of the Turkish Version of the Appetite Loss in Older Adults With and Without Cognitive Impairment (ALOC) Screening Scale | From enrollment to the end of treatment at 12 weeks
  Loss of appetite is common in older adults and increases the risk of malnutrition, functional decline, and adverse health outcomes. Older adults with cognitive impairment are particularly vulnerable. The Appetite Loss in Older Adults With and Without Cognitive Impairment (ALOC) Screening Scale, developed by Rudzinska et al. (2025), consists of 7 dichotomous items scored 0-7, with cut-offs indicating appetite loss (≥3), risk (=2), or low risk (≤1). This study aims to adapt the ALOC into Turkish and evaluate its psychometric properties in adults ≥65 years with and without cognitive impairment. Internal consistency, test-retest reliability, factor structure, convergent and known-groups validity, and diagnostic accuracy will be tested. Predictive validity will be assessed through nutritional and clinical outcomes over 3 months. The validated Turkish ALOC is expected to provide a practical screening tool to support early detection and management of appetite loss in geriatric care.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin Aid and Kindness Foundation Retirement Home, Mersin Sevgi Bağı Retirement Home, Private Mersin Bahar Retirement Home and Private Alya Elderly Care Center and Retirement Home., Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No